CLINICAL TRIAL: NCT00314899
Title: Fetal Immunity to Plasmodium Falciparum Malaria
Brief Title: Fetal Immunity to Falciparum Malaria
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0074
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2009-04

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria, Plasmodium falciparum, Kenya, immunity
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The purpose of this study is to find out what effect malaria in the mother has on the development of her child's immune system response to malaria and whether being exposed to malaria in the womb makes a child more likely to get malaria. The study will also assess the effect that exposure to malaria in the womb has on the child's growth and development over the first three years of life. Study participants will include 480 healthy pregnant women (greater than or equal to 15 years of age), their healthy offspring, 20 healthy people from the United States with no malaria exposure or disease and 40 adult Kenyans who have previously been exposed to malaria or have malaria with no signs of infection. Study procedures will include an ultrasound (procedure to assess the baby's growth and development in the womb), blood, urine, and stool collections. Newborns will be examined at birth, and at 6, 12, 18, 24, 30 and 36 months of age.

DETAILED DESCRIPTION:
The primary aim of this study is to determine how prenatal exposure to malaria influences development of humoral and cellular immune responses to malaria blood stage antigens from birth to 3 years of age. In addition, the study will determine the risk factors and mechanisms associated with congenital malaria or exposure of the fetus to malaria blood stage antigens, assess how prenatal exposure to malaria affects susceptibility to malaria infection during infancy, and evaluate how perinatal exposure to malaria affects growth and development during infancy. A primary goal of this research will be to examine a cohort of infants from birth to 36 months of age; the predictive value of allele-specific invasion inhibitory antibodies to Merozoite Surface Protein 1 (MSP1) and antibody titers to MSP1 will be evaluated with respect to type and magnitude of neonatal cellular and humoral immune response to MSP1. An understanding of natural immunity to MSP1, and the influence of prenatal exposure, may be critical to informed interpretation of immunologic, parasitologic, and clinical endpoints of vaccine trials using blood stage antigens that will be ultimately directed to infants and children. Healthy adult pregnant women (greater than or equal to 15 years of age) and their healthy offspring (beginning at birth) will be followed until they are 36 months old. Newborns will be examined at birth and at 6, 12, 18, 24, 30 and 36 months of age. Enrollment will occur at time of first visit to the antenatal clinic during the second trimester when peripheral blood, stool, and urine samples will be obtained from each pregnant woman. A finger stick blood sample will be obtained from the mothers at each subsequent antenatal visit to assess the presence of malaria during pregnancy. An ultrasound examination will be done on the mothers at the initial antenatal visit to assess gestational age and at 26-30 weeks to assure proper growth and development of fetus and to screen for any potential problems. At delivery venous and finger stick blood, stool, and urine will be obtained from the mother. Umbilical cord and placental blood, and a placental biopsy will be obtained, and thereafter infants will be followed every 6 months (plus or minus 2 months). A physical examination of infants will be done and peripheral blood, stool, and urine will be obtained from infants. The study population will also include about 20 healthy adult North American control subjects with no malaria exposure or infection and about 40 adult Kenyans who either have been exposed to malaria or have asymptomatic malaria infection.

ELIGIBILITY:
Inclusion Criteria:

* At least greater than or equal to 15 years of age.
* Willingness to provide informed consent.
* Confirmed pregnancy.
* Apparent good health.
* Long-term residence in Msambweni locations who anticipate residing in the area during the study period (at least 3 years). Women whose immediate and/or extended families do not reside in Kwale District will be discouraged from enrolling in the study.
* Willingness to donate blood (peripheral venous blood or fingerstick blood as per the protocol) during ANC visits and at the time of delivery.
* Willingness to release human immunodeficiency virus (HIV) testing results from the voluntary counseling and treatment (VCT) program, or be tested by our staff and, if positive, to have their infants tested for HIV at 12 and 24 months of age.
* Willingness of the infant's mother to participate in prenatal and postnatal care at Msambweni District Hospital.
* Willingness of the mother/caregivers to participate in a prospective survey that involves bi-annual venipuncture (3-5 mL blood volume) of the infant commencing at 6 months (plus or minus 2 months of age) and ending at age 36 months.
* Multiple births can be included.

Pregnant women will be allowed to enroll irrespective of their gestational age, although they cannot enroll at delivery because they cannot undergo adequate consent. However, potential participants will be strongly encouraged to come to the clinic for prenatal care early in the second trimester (ideally <16 weeks gestation) both to ensure adequate prenatal care for the mother and unborn infant and to provide sufficient follow-up time to collect multiple antenatal study samples from the mother.

Inclusion criteria for American participants: Participants must be in good health, between the ages of 18 to 65, and have never been exposed to malaria.

Inclusion criteria for Kenyan control subjects: Participants must be in general good health and either have been exposed to malaria or be infected with malaria, but asymptomatic. Exposure will be determined by the presence of antibodies to malarial blood-stage antigens, eg, MSP1-42. Subjects must be aged 18 to 55 years, inclusive.

Exclusion Criteria:

* Preterm delivery less than 34 weeks gestation.
* Failure to deliver in the hospital.
* Evidence of placenta previa.
* Maternal chorioamnionitis.
* Receipt of immunosuppressive drugs during pregnancy.
* Hemoglobin less than 6.07 g/dL for females*.
* More One plus or greater glucose in urine.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding enrollment in the study.
* Simultaneous participation in any other interventional clinical trial.
* Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, or any other findings that in the opinion of the CO or PI may increase the risk of participating in the study.
* Other conditions that in the opinion of the CO or PI would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol.

  * These values may change base on survey of adult normal laboratory test values in Msambweni. Values for children will be revised based on a survey of pediatric normal values in Msambweni.

Censoring events for the mother and newborn (and, by default, the infant's mother):

* Mother delivers elsewhere, migrates out of area, dies, spontaneous abortion or stillbirth.
* APGAR score for the infant of less than 5 at 10 minutes after birth.
* Muconium aspiration, respiratory distress syndrome, or condition to require neonatal resuscitation.
* Extremely low birth weight (less than 1500 grams).
* Refuse to continue to participate in the study.

Participants who move outside the study area during the course of the study will be dropped from further participation. However, data collected to that point may be included in analysis.

Exclusion of American and Kenyan control subjects:

No prior screening will be performed for the American control subjects, other than that they state they are healthy and have no acute or chronic medical problems. For the Kenyan adult control subjects, they will also be queried about their general overall perceived health and will have no known acute or chronic illnesses. A FSB sample will be obtained from the Kenyan control subjects and tested for anti-bodies to MSP142, a blood smear for malaria, and hemoglobin concentration by Hemacue test. If the hemoglobin concentration is <10 gm/dL, the subject will not be asked to donate blood and will be referred to the appropriate health care deliverers to receive appropriate treatment (oral iron supplements).

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-09-15; Primary Completion 2009-11-15 (Actual); Study Completion 2010-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI Centre for Geographic Medicine Research, Nairobi, Kenya